CLINICAL TRIAL: NCT01956747
Title: Optimization of Systemic Treatment Strategies in Elderly Patients With Advanced Solid Malignancies
Acronym: OptiMal
Status: Completed | Type: Observational
Sponsor: Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, K. Versteeg, Medical Oncologist, Amsterdam UMC, location VUmc
Other Study IDs: 2013/164
Record Dates: First submitted 2013-09-27; First posted 2013-10-08 (Estimated); Last update posted 2020-11-20 (Actual); Status verified 2020-11

CONDITIONS: Colorectum Advanced Malignancies; Breast Advanced Malignancies; Prostate Advanced Malignancies

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- standard anticancer treatment: Patients older than 70 years of age with advanced malignancies of colorectum, breast or prostate, who will start with full standard anticancer treatment as decided by their oncologist.
  Interventions: Procedure: venapunction; Procedure: bone marrow punction

INTERVENTIONS:
Procedure: venapunction
Procedure: bone marrow punction

SUMMARY:
The purpose of this study is to assess whether the presence of a Myelodysplastic Syndrome (MDS) , Idiopathic Cytopenia of Undetermined Significance (ICUS) or Idiopathic Dysplasia of Undetermined Significance (IDUS), correlates with treatment intensity and clinical outcome in older patients with advanced malignancies receiving palliative chemotherapy. We will study the relation between sarcopenia, comprehensive geriatric assessment en pharmacokinetics with treatment related toxicity as well. We hypothesize that a standardized flow cytometry test to determine bone marrow capacity, a Comprehensive Geriatric Assessment and/or measurement of human body composition with computerized tomography will provide an accurate tool to optimize treatment strategies in elderly patients with advanced malignancies.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 70 years
* Diagnosis of advanced cancer of colorectum, breast or prostate
* Standard first line palliative treatment with cytotoxic agents will be started (Folfox, Xelox, capecitabine, paclitaxel or docetaxel)
* Estimated life expectancy ≥ 3 months
* Able to give informed consent
* WHO performance status ≤ 2
* Absence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the treatment and follow-up schedule; those conditions should be assessed with the patient before registration in the trial
* No other severe medical or psychiatric conditions that in the judgment of the investigator renders the patient inappropriate for inclusion in this study.
* Before patient registration, written informed consent must be given and documented to ICH/EUCGCP, national/local regulatory requirements and the local rules followed in our institution

Exclusion Criteria:

* Presence of cytopenia due to iron-, vitamin B12 and folic acid deficiency or hemolysis, unless adequately supplemented.
* Creatinine clearance ≤ 30 ml/min
* Serum AST and ALT ≥ 2.5 x ULN, in case of liver metastases serum AST and ALT ≥ 5 x ULN
* In case of therapy with Docetaxel/Paclitaxel serum bilirubin ≥ 1.5 x ULN

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients older than 70 years of age with advanced malignancies of colorectum, breast or prostate, who will start with full standard anticancer treatment as decided by their oncologist
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2013-07; Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
To determine whether the presence of a low - intermediate 1 risk MDS, IDUS or ICUS can predict for (myelo)toxicity in older patients with advanced malignancies receiving palliative chemotherapy | from date of study inclusion until 30 days after end of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- VU Medical Center, Amsterdam, Netherlands